CLINICAL TRIAL: NCT06664203
Title: Comparison of the Anesthetic and Analgesic Efficacy of Selective Truncal Blocks at Different Volumes in Upper Extremity Orthopedic Surgeries
Brief Title: Efficacy of Variable Volume Truncal Blocks in Upper Limb Orthopedic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SERPİL ŞEHİRLİOĞLU, principal invertigator, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaTREH-SeTb
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Pain Management; Anaesthesia Complication
Keywords: postoperative pain; selective turuncus block; arm anaesthesia
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with 15 ml SeTb group (Active Comparator): This group will receive a SeTB (Selective Trunk Block) with a total of 15 ml of bupivacaine
  Interventions: Procedure: Selective turuncus block with 15 ml bupivacain
- With 25 ml bupivacain SeTb (Active Comparator): This group will receive a SeTB (Selective Trunk Block) with a total of 25 ml of bupivacaine
  Interventions: Procedure: Selective turuncus block with 25 ml bupivacain

INTERVENTIONS:
Procedure: Selective turuncus block with 25 ml bupivacain — A high-frequency linear ultrasound (USG) probe will be used to locate the C7 transverse process, which will serve as a sonoanatomic landmark. Once the C5 ventral ramus is identified at the C7 transverse process level, the linear probe will be slightly caudally angled to visualize the C6 ventral ramus. The area where the superior trunk is formed by C5 and C6 will be examined with the USG probe until the superior trunk is visualized. Below the superior trunk, the middle trunk and the C8 ventral ramus will be visible. In Group 1, a total of 23 ml of 0.5% bupivacaine plus 2 ml (8 mg dexamethasone) will be used as the local anesthetic mixture, totaling 25ml. 7ml of the local anesthetic mixture will be injected into the superior trunk, the middle trunk for an additional 8 ml. The probe will then be directed caudally to obtain an optimal view of the lower trunk, where 10 ml of the same mixture will be injected close to the lower trunk.
  Arms: With 25 ml bupivacain SeTb
Procedure: Selective turuncus block with 15 ml bupivacain — In Group 2, 13 ml of 0.5% bupivacaine plus 2 ml (8 mg dexamethasone) will be used, totaling 15 ml. In Group 2, 5 ml of the local anesthetic mixture will be injected into the superior trunk, followed by 5 ml into the middle trunk and 5 ml into the lower trunk, as in Group II.
  Arms: with 15 ml SeTb group

SUMMARY:
aim of this study is to compare the effect of selective truncal blocks, performed at different doses and volumes, on the onset times of motor and sensory blocks required for anesthesia in patients scheduled for hand, wrist, forearm, and elbow surgeries. Completing the operation under regional anesthesia will be considered a successful block.

DETAILED DESCRIPTION:
The primary outcome of this study is to compare the effect of selective truncal blocks, performed at different doses and volumes, on the onset times of motor and sensory blocks required for anesthesia in patients scheduled for hand, wrist, forearm, and elbow surgeries. Completing the operation under regional anesthesia will be considered a successful block.

Secondary Outcome Variables:

Secondary outcomes include comparisons between the two groups regarding total motor block duration and analgesia durations, tourniquet pain, incidence of diaphragm paralysis, complications (vascular puncture, paresthesia, Horner's syndrome, hoarseness), time to first postoperative analgesic administration, and total analgesic consumption within the first 24 postoperative hours.

This study aims to compare the anesthetic efficacy and complication rates associated with different volumes of local anesthetic used in upper extremity surgeries (elbow, forearm, and hand surgeries) in patients over 18 years of age with ASA scores of 1-2 to reduce complication rates.

In recent years, brachial plexus blocks, performed through various approaches, have become preferred over general anesthesia for upper extremity surgeries due to numerous advantages. Peripheral nerve blocks are known to maintain patient consciousness and spontaneous breathing, reduce airway interventions, provide effective postoperative pain control, decrease opioid-related side effects, limit surgical stress-induced metabolic and endocrine changes, enable early discharge, and reduce treatment costs.

The selective truncal block approach has rapid onset and high success rates. The use of ultrasound guidance in peripheral blocks has also reduced various complications, such as vascular injury. The selective truncal approach, defined by Manoj Kumar Karmakar in 2020, involves blocking the upper, middle, and lower trunks of the brachial plexus at the C7 transverse process level, achieving sensory and motor blockade across all ipsilateral upper extremity dermatomes except T2. Interscalene block, which targets the roots of the brachial plexus, may lead to complications such as Horner's syndrome and ipsilateral diaphragm paralysis due to phrenic nerve blockade. This study aims to compare the efficacy and complications of truncal blocks applied at different volumes in the selective truncal approach at the trunk level, reducing complications such as phrenic nerve paralysis and Horner's syndrome.

Higher volumes of local anesthetics are associated with increased complication risks, whereas lower volumes may result in block failure. The adjuvant use of dexamethasone allows for more effective anesthetic and analgesic efficacy at lower volumes and aims to reduce complications such as phrenic nerve paralysis and Horner's syndrome. Given the potential spread of high local anesthetic volumes to the phrenic nerve, 8 mg of dexamethasone will be added to both groups to facilitate lower volume usage.

Dexamethasone is a widely used glucocorticoid with anti-inflammatory and anti-toxic effects, characterized by potent lipophilic activity. It is fat-soluble and increases pH, facilitating the penetration of local anesthetics into the nerve sheath, and has been shown to prolong the duration of action of local anesthetics. Additionally, dexamethasone is commonly used in pain management due to its neuromodulatory effects.The selective trunk block targets the trunks of the brachial plexus, blocking the nerves at the trunk level rather than the root level. Today, the brachial plexus block is often preferred over general anesthesia in upper extremity surgeries due to several advantages, such as preservation of consciousness, minimized respiratory impact, reduced airway intervention, long-lasting postoperative pain control, fewer opioid-related side effects, limited metabolic and endocrine changes associated with surgery, and early discharge. In interscalene brachial plexus blocks, diaphragm paralysis and Horner syndrome are common due to the proximity to the phrenic nerve. In infraclavicular and supraclavicular blocks, the close proximity to the pleura presents a disadvantage; however, the widespread use of ultrasound guidance has reduced the risk of complications associated with this proximity. In 2020, Manoj Kumar Karmakar introduced the selective trunk approach, suggesting that blocking the upper, middle, and lower trunks of the brachial plexus at the C7 transverse process level produces sensory and motor blocks in all ipsilateral upper extremity dermatomes except T2. However, diaphragm paralysis and Horner syndrome can still occur with high-volume local anesthetic applications at this level.

This study aims to compare the anesthetic efficacy and complication rates of selective trunk blocks with different volumes. After informed consent is obtained, all patients will be taken to the preoperative intervention room 40 minutes before surgery for the block application. Both groups will receive a selective trunk block. An IV line will be placed for each patient, who will be monitored and given 0.05 mg/kg IV midazolam for sedation.

Patients will be randomized into two groups using a sealed envelope method. Group 1 will receive a selective trunk approach peripheral nerve block with a volume of 25 ml, and Group 2 will receive a volume of 15 ml. Different anesthesiologists will administer the block and perform postoperative follow-ups.

Patients will be placed in a supine position without a pillow, with arms aligned alongside the body and the head turned away from the block side. A high-frequency linear ultrasound (USG) probe will be used to locate the C7 transverse process, which will serve as a sonoanatomic landmark. Once the C5 ventral ramus is identified at the C7 transverse process level, the linear probe will be slightly caudally angled to visualize the C6 ventral ramus. The area where the superior trunk is formed by C5 and C6 will be examined with the USG probe until the superior trunk is visualized. Below the superior trunk, the middle trunk and the C8 ventral ramus will be visible. The T1 ventral ramus will be seen on the first rib upon caudal angling of the probe. After obtaining all these images, the block needle will be directed from lateral to medial. In Group 1, a total of 23 ml of 0.5% bupivacaine plus 2 ml (8 mg dexamethasone) will be used as the local anesthetic mixture, totaling 25 ml. In Group 2, 13 ml of 0.5% bupivacaine plus 2 ml (8 mg dexamethasone) will be used, totaling 15 ml. In Group 1, 7 ml of the local anesthetic mixture will be injected into the superior trunk, and the needle will then be slightly withdrawn and redirected to the middle trunk for an additional 8 ml. The probe will then be directed caudally to obtain an optimal view of the lower trunk, where 10 ml of the same mixture will be injected close to the lower trunk. In Group 2, 5 ml of the local anesthetic mixture will be injected into the superior trunk, followed by 5 ml into the middle trunk and 5 ml into the lower trunk, as in Group 1.

After the block is performed, sensory and motor blocks in the median, ulnar, radial, musculocutaneous, and axillary nerve dermatomes will be assessed every 10 minutes for 30 minutes. Sensory block will be evaluated using the pinprick test (0: no sensory block, 1: touch sensation but no pain, 2: no touch or pain sensation). For the block to be considered sufficient for anesthesia, the following criteria must be met:

Sensory block level of 1 in all dermatomes at 30 minutes. Motor block in at least three of the musculocutaneous, radial, ulnar, median, and axillary nerves.

If there is no motor block in three or more distal peripheral nerves, general anesthesia will be administered, and the patient will be excluded from the study. Diaphragm thickening fractions during expiration and deep inspiration will be measured with ultrasound before and 30 minutes after the block to evaluate diaphragm paralysis. All patients will be monitored for Horner syndrome. Once in the operating room, all patients will receive midazolam at 0.4 - 0.5 mg/kg IV to maintain a Ramsey sedation scale of 3-4.

Pain will be assessed intraoperatively using the Visual Analog Scale (VAS). If VAS ≥3, the patient will initially receive a 0.1 mcg/kg IV bolus of fentanyl. If the VAS remains ≥3 after 15 minutes, an additional 0.1 mcg/kg fentanyl dose will be administered. If the VAS remains ≥3 after these interventions, general anesthesia will be administered, and the block will be considered unsuccessful.

Patients will be assessed postoperatively for motor block and analgesic efficacy at 2, 4, 8, 12, and 24 hours, with VAS tracking. The postoperative assessments will be conducted by an observer blinded to the block administration. Motor block will be considered resolved once motor function returns in two or more nerves (median, musculocutaneous, radial, ulnar, axillary). Analgesic efficacy will be considered resolved if VAS >3. For rescue analgesia, 1 gram of paracetamol IV will be administered, with an additional 1 mg/kg tramadol if pain persists after 15 minutes.

The time to achieve sensory block in all dermatomes after the block will be recorded as the "ready for surgery" time. Intraoperative tourniquet pain records will be kept. The time to first postoperative analgesic use and total analgesic consumption within 24 hours postoperatively will be recorded, and patients will be evaluated for complications.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Body Mass Index (BMI) of 18-35 kg/m²
* Age: 18-65 years -Patients undergoing all upper extremity orthopedic surgeries, except shoulder surgeries (distal humerus, elbow, forearm, hand, and wrist), will be included. -

Exclusion Criteria:

* Patient refusal
* Pregnancy or breastfeeding
* Severe pulmonary disease
* Contralateral diaphragm paralysis
* Nerve injury secondary to trauma
* Neuromuscular disease
* Peripheral neuropathy
* Bleeding diathesis
* Allergy to local anesthetics and dexamethasone
* Uncontrolled diabetes mellitus
* Morbid obesity with BMI >35
* Severe cardiovascular, renal, or hepatic disease
* Infection at the site of the nerve block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
on the onset times of motor and sensory blocks required for anesthesia | 24 hour
  The primary outcome of this study is to compare the effect of selective truncal blocks, performed at different doses and volumes, on the onset times of motor and sensory blocks required for anesthesia in patients scheduled for hand, wrist, forearm, and elbow surgeries. Completing the operation under regional anesthesia will be considered a successful block.

SECONDARY OUTCOMES:
Total Opioid Consumption | 24 hour
  total analgesic consumption within the first 24 postoperative hours
time to first rescue analgesic requirement. | 24 hour
  time to first postoperative analgesic administration,
diaphragm paralysis | 24 hour
  ASSESMENT OF diaphragm paralysis

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Sehirlioglu, MD, Principal Investigator — Gaziosmanpasa Research and Training Hospital
Locations (1):
- Gaziosmanpasa Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data associated with the paper are not publicly available but are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: FİRST 5 YEARS
Access Criteria: drserpilsahin@gmail.com

REFERENCES:
- [Result] Sivashanmugam T, Sripriya R, John Paul S, Ravishankar M. Estimation of minimum effective local anaesthetic volume to block the lower trunk during selective truncal injection brachial plexus block. Indian J Anaesth. 2022 Aug;66(Suppl 5):S281-S283. doi: 10.4103/ija.ija_1087_21. Epub 2022 Aug 12. No abstract available. PMID 36262721
- [Result] Bao X, Huang J, Feng H, Qian Y, Wang Y, Zhang Q, Hu H, Wang X. Effect of local anesthetic volume (20 mL vs 30 mL ropivacaine) on electromyography of the diaphragm and pulmonary function after ultrasound-guided supraclavicular brachial plexus block: a randomized controlled trial. Reg Anesth Pain Med. 2019 Jan;44(1):69-75. doi: 10.1136/rapm-2018-000014. PMID 30640655